CLINICAL TRIAL: NCT05804591
Title: The Effect of Preemptive Oral Pregabalin As an Element of Multimodal Analgesia in Patients Undergoing Laparoscopic Sleeve Gastrectomy. a Randomized, Prospective, Double Blind Study.
Brief Title: Pregabalin in the Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy (LSG).
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PreGab LSG
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Postoperative Pain; Postoperative Nausea and Vomiting; Opioid Use
Keywords: Laparoscopic sleeve gastrectomy; Obesity; Pregabalin; Multimodal analgesia
MeSH Terms: conditions — Obesity; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal analgesia group (Placebo Comparator): Patients receiving placebo per os 1 hour preoperatively and anesthesia with standard, multimodal analgesia afterwards.
  Interventions: Drug: Placebo
- Multimodal analgesia with preemptive pregabalin group (Experimental): Patients receiving pregabalin 150mg per os 1 hour preoperatively and anesthesia with standard, multimodal analgesia afterwards.
  Interventions: Drug: Pregabalin 150mg

INTERVENTIONS:
Drug: Pregabalin 150mg — Single dose of pregabalin 150mg in a capsule per os 1 hour before start of the operation.
  Arms: Multimodal analgesia with preemptive pregabalin group
Drug: Placebo — 1 capsule containing placebo per os 1 hour before start of the operation.
  Arms: Multimodal analgesia group

SUMMARY:
The aim of this clinical trial is to assess preemptive oral pregabalin administration in the obese patients undergoing laparoscopic sleeve gastrectomy. The main aims of the study are to evaluate postoperative pain treatment and effect on the intraoperative hemodynamical stability.

The participants will be divided into 2 groups: with or without preemptive pregabalin administration.

DETAILED DESCRIPTION:
Pregabalin is a GABA analogue that has analgesic, anxiolytic and effects. There are studies indicating that this drug can be used as an element of multimodal analgesia to decrease opioid requirements in postoperative period. Such an effect would be particularly beneficial for patients with obesity scheduled for laparoscopic sleeve gastrectomy, most commonly performed bariatric surgery.

The investigators hypothesized that preemptive pregabalin administration may improve quality of postoperative pain score with less incidence of opioid side effects as well as similar or better intraoperative hemodynamical stability.

ELIGIBILITY:
Inclusion Criteria:

* Sleeve gastrectomy in patients with BMI > 40 or >35 with comorbidities
* Written informed consent

Exclusion Criteria:

* Patient's refusal
* Known allergies to study medication
* Inability to comprehend or participate In pain scoring scale
* Inability to use intravenous patient controlled analgesia
* Changes of operation extent during procedure
* Revisional operations
* End stage organ failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Total postoperative oxycodone consumption | Day "0"
  PCA (Patient's controlled analgesia) iv pump, oxycodone will be administered on patient's demand by 2mg boli, with lock out time 10 minutes
Postoperative pain score in NRS scale | Day "0", assessed 1 hour after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable
Postoperative pain score in NRS scale | Day "0", assessed 6 hour after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable
Postoperative pain score in NRS scale | Day "0", assessed 12 hour after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable
Postoperative pain score in NRS scale | Day "0", assessed 24 hour after operation
  NRS range from 0 for no pain to 10 for worst pain imaginable

SECONDARY OUTCOMES:
Postoperative sedation score | Day "0", assessed 1,6,12 and 24 hours after operation
  1-6 Ramsay sedation score; 1 - agitated or restless 6 - unresponsive
Postoperative nausea and vomiting | Day "0", assessed 1,6,12 and 24 hours after operation
  Simplified PONV impact scale 0-6 0 - no nausea nor vomiting 6 - >3 episodes of vomiting and nausea all of the time
Highest BP | intraoperative
  Highest BP during operation
Lowest BP | intraoperative
  Lowest BP during operation
Highest HR | intraoperative
  Highest HR during operation
Lowest HR | intraoperative
  Lowest HR during operation
Total ephedrine dosis | intraoperative
  Ephedrine is a vasopressor used in case of hypotension to maintain mean arterial pressure > 65 mmHg or to increase blood pressure to check surgical hemostasis
Postoperative desaturation | Day "0", assessed 1,6,12 and 24 hours after operation
  SpO2 < 94%
Blurred vision | Day "0", assessed 1,6,12 and 24 hours after operation
  Presence of blurred or abnormal vision
Patient's comfort assessed in QoR-40 formulary | Day "0", assessed 24 hours after operation
  QoR-40 (Quality of Recovery) scale is used to measure the quality of recovery after surgery and anesthesia, it is a 40 item questionnaire that provides a score across five dimensions: patient support, comfort, emotions, physical independence, and pain. Formulary will assess first 24 hours following the operation. Maximal score is 200, higher result is associated with better quality of recovery.
Postoperative oxycodone consumption | Day "0", assessed 1,6,12 and 24 hours after operation
  PCA (Patient's controlled analgesia) iv pump, oxycodone will be administered on patient's demand by 2mg boli, with lock out time 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Mieszczański, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Szpital Kliniczny Dzieciatka Jezus, Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mieszczanski P, Gorniewski G, Janiak M, Trzebicki J. The effect of pre-emptive oral pregabalin on opioid consumption in patients undergoing laparoscopic sleeve gastrectomy with an analysis of intraoperative hemodynamic stability and quality of recovery: study protocol for a randomized, prospective, double-blind study. Trials. 2024 Jun 7;25(1):367. doi: 10.1186/s13063-024-08225-3. PMID 38849875